CLINICAL TRIAL: NCT04055207
Title: VA Video Connect to Improve Access to Multi-disciplinary Specialty Care
Brief Title: VA Video Connect in HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 18-077; I01HX002645 (NIH)
Record Dates: First submitted 2019-07-24; First posted 2019-08-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: HIV
Keywords: HIV; Telemedicine

STUDY DESIGN:
Intervention Model Description: Veterans in the Infections Disease clinic at the Michael E. DeBakey Veterans Affairs Medical Center (MEDVAMC) will be randomly assigned to either an offer of VA Video Connect (VVC) delivered HIV care or to usual care for HIV. All treatment as usual options for HIV care will be available to all patients in both treatment arms, however only the Veterans in the VVC arm will be actively offered this VA-approved technology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VVC (Experimental): Option to receive VA Video Connect (VVC) delivery of HIV care.
  Interventions: Other: VVC
- Usual Care (No Intervention): All HIV care available at MEDVAMC will be delivered as usual.

INTERVENTIONS:
Other: VVC — Telehealth treatment is delivered via VA-approved technology to a patient's computer or mobile device.
  Other Names: VA Video Connect
  Arms: VVC

SUMMARY:
The purpose of this research study is to see how effective the addition of video to home telehealth services is in helping patients with HIV to remain in care, which is vital to management of their illness. The investigators also want to understand how to best put the video to home services into practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the Infectious Diseases clinic at Michael E. DeBakey VA Medical Center (MEDVAMC), Houston, TX, with HIV infection
* At least 18 years of age
* Able to speak English
* Able to consent to the use of VVC

Exclusion Criteria:

* Unable to use or consent to use VVC, due to either significant physical or mental disability
* Incarcerated (though MEDVAMC does not generally provide care for prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Constancy retention in care measure | 12 months
  Percentage of patients who completed at least 1 visit with a primary care or Infectious Diseases provider in each 6 months of the year at least 60 days apart.

SECONDARY OUTCOMES:
Adherence retention in care measure | 12 months
  Percentage of scheduled HIV clinic appointments attended over the year
Completed visits for adherence counseling | 12 months
  Number of completed visits for counseling, mental health, and social services during the year.
HIV suppression | 12 months
  Percentage of Veterans with HIV on ART whose most recent viral load during the 12-month period was <200c/mL
Adherence to ART medications | 12 months
  Number of ART medication pills dispensed from pharmacy over the year divided by days in year.

OTHER OUTCOMES:
AUDIT | 12 months
  10-item screening tool to assess alcohol consumption, drinking behaviors and alcohol-related problems. Item responses range from 0-4. Scores range from 0-40. Higher scores indicate more harmful alcohol use.
Patient Health Questionnaire depression scale (PHQ-9) | 12 months
  Brief measure of depression symptoms consisting of 9 items rated from 0-3 (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). Scores range from 0 to 27. Higher scores indicate greater depression severity.
Posttraumatic Disorder Checklist (PCL-5) total | 12 months
  Measure of PTSD symptoms. 20 items rated from 0 (not at all) to 4 (extremely). Scores range from 0 to 80. Higher scores = higher symptom severity.
Montreal Cognitive Assessment (MoCA) | 12 months
  Brief screening tool that assesses cognitive functioning across 8 domains; attention and concentration, executive functions, memory, language, conceptual thinking, calculations and orientation. Scores range from 0-30. Higher scores indicate greater cognitive function.
CD4 cell count | 12 months
  Last recorded value in medical record during 12 month period
HIV viral load | 12 months
  Last recorded value in 12 months period.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Alexandra Lindsay, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson JL, Matchanova A, Beltran-Najera I, Ridgely NC, Mustafa A, Babicz MA, Hasbun R, Giordano TP, Woods SP. Preliminary Validity of a Telephone-Based Neuropsychological Battery in a Consecutive Series of Persons with HIV Disease Referred for Clinical Evaluation. Arch Clin Neuropsychol. 2023 May 22;38(4):570-585. doi: 10.1093/arclin/acac104. PMID 36566509
- [Background] Sheinfil AZ, Day G, Walder A, Hogan J, Giordano TP, Lindsay J, Ecker A. Rural Veterans with HIV and Alcohol Use Disorder receive less video telehealth than urban Veterans. J Rural Health. 2024 Jun;40(3):419-429. doi: 10.1111/jrh.12799. Epub 2023 Sep 27. PMID 37759376
- [Derived] Gloston GF, Day GA, Touchett HN, Marchant-Miros KE, Hogan JB, Chen PV, Amspoker AB, Fletcher TL, Giordano TP, Lindsay JA. Pivoting to Video Telehealth for Delivery of HIV Care During COVID-19: A Brief Report. Telemed Rep. 2021 Aug 6;2(1):205-210. doi: 10.1089/tmr.2021.0010. eCollection 2021. PMID 34841420

DOCUMENTS (1):
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT04055207/ICF_000.pdf